CLINICAL TRIAL: NCT02365467
Title: Evaluation of the Valiant Mona LSA Thoracic Stent Graft System in Descending Thoracic Aortic Aneurysms and Chronic Dissections
Brief Title: Evaluation of the Valiant Mona LSA Thoracic Stent Graft System in Descending TAA and Chronic Dissections
Status: Completed | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10151194DOC
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Results first posted 2022-10-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Aortic Aneurysm, Thoracic, Chronic Type B Dissection
Keywords: TEVAR; Thoracic Aneurysm; Endovascular Aortic Repair; Type B Dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with Valiant Mona LSA device (Experimental): Treatment with Valiant Mona LSA device
  Interventions: Device: Valiant Mona LSA Thoracic Stent Graft System

INTERVENTIONS:
Device: Valiant Mona LSA Thoracic Stent Graft System

SUMMARY:
The purpose of the Feasibility study is to characterize the safety of the Valiant Mona LSA Thoracic Stent Graft System, including an assessment of the safety and effectiveness of the device acutely and at the 30 day visit in the identified subject population. This study will also evaluate the current instructions for use and may direct changes to the delivery and deployment steps.

The purpose of the expansion to the Feasibility Study is to characterize the Valiant Mona LSA Thoracic Stent Graft System, in particular to assess the safety and effectiveness of the device acutely and at the 30 day visit, in subjects enrolled with chronic, Type B dissections.

DETAILED DESCRIPTION:
The purpose of the clinical investigation is to assess the feasibility of the Valiant Mona LSA Thoracic Stent Graft System to repair fusiform/saccular aneurysms, penetrating ulcers and chronic type B dissections of the DTA in patients who require coverage of the LSA, including an assessment of the safety and effectiveness of the device acutely and at the 30 day visit in the identified subject population. Procedural information will be collected in order to enhance the current instructions for use and delivery and deployment steps.

The chronic Type B Dissection expansion subjects will be prospectively enrolled in support of a future premarket approval analysis for the Valiant Mona LSA device.

ELIGIBILITY:
Inclusion Criteria for Thoracic Aortic Aneurysms and Penetrating Ulcers:

* Subject is at least 18 years of age.
* Subject understands and has signed an Informed Consent approved by the Sponsor and by the IRB for this study.
* Subject must be considered a candidate for revascularization of the LSA. Subject must be able to tolerate a surgical revascularization of the LSA.
* Subject has a TAA/PAU which will require coverage of the LSA and is:

  * a fusiform aneurysm with a diameter of ≥ 5.5 cm OR is > 2 times the diameter of the non-aneurysmal thoracic aorta; AND/OR
  * a saccular aneurysm or PAU (ulcer defined as ≥ 10 mm in depth and 20 mm in diameter, or symptomatic)
* Subject has a healthy, non-diseased aortic proximal seal zone of at least 20 mm from the distal end of the LCC ostium to the beginning of the disease, including at least 10 mm between the LSA and the LCC.
* Subject has a non -diseased aortic proximal neck length of >0mm distal to the LSA
* Subject has a non-diseased aortic diameter between 25 mm and 42 mm
* Subject has a non-diseased LSA with a diameter between 8 mm and 13 mm.
* Subject has sufficient landing zone within the LSA to accommodate the BSG without occlusion of any significant vessels
* Brachial, iliac or femoral artery access vessel morphology (diameter, calcification, tortuosity) that is compatible with vascular access techniques, the device, or accessories.

  * Introducer sheath is required for all procedures.
  * An iliac conduit is required for access if the above requirements are not met.

Inclusion Criteria for Chronic Type B Dissections:

* Subject is at least 18 years of age.
* Subject understands and has signed an Informed Consent approved by the Sponsor and by the IRB for this study.
* Subject must be considered a candidate for revascularization of the Left Subclavian Artery (LSA). Subject must be able to tolerate a surgical revascularization of the LSA.
* Subject has a chronic type B dissection which will require coverage of the LSA. A chronic type B dissection is defined as > 30 days from symptom onset and is complicated with an aortic diameter ≥ 5.5 cm or has progressive aortic enlargement (> 5 mm/year).
* Subject has a healthy, non-diseased aortic proximal seal zone of at least 20 mm from the distal end of the LCC ostium to the beginning of the disease, including at least 10 mm between the LSA and the LCC
* Subject has a non-diseased aortic diameter between 28 mm to 44 mm.
* Subject has a non-diseased LSA with a diameter between 8 mm and 13 mm.
* Subject has sufficient landing zone within the LSA to accommodate the BSG without occlusion of any significant vessels
* Brachial, iliac or femoral artery access vessel morphology (diameter, calcification, tortuosity) that is compatible with vascular access techniques, the device, or accessories.

  * Introducer sheath is required for all procedures.
  * An iliac conduit is required for access if these requirements are not met.

Exclusion Criteria

* Subjects will be excluded if they have conditions requiring prospective revascularization of the LSA including:

  * Dominant left vertebral artery requiring revascularization
  * Prior coronary artery bypass graft utilizing the left mammary artery requiring revascularization
  * Incomplete circle of Willis or other neurological vasculature requiring revascularization
* Subject has an aneurysmal, tortuous, or atherosclerotic LSA.
* Subject has an acute dissection of the descending thoracic aorta.
* Subject has an intramural hematoma of the descending thoracic aorta.
* Subject has prohibitive calcification, occlusive disease, or tortuosity of intended fixation sites.
* Subject has circumferential calcification in the external iliac artery or in the common iliac artery with an intraluminal diameter (ID) less than 10mm at any point proximal to or at the access vessel site unless a surgical adjunctive procedure is planned.
* Subject requiring an aortic conduit or direct aortic access
* Subject has an aortic atheroma classified as grade IV or grade V.
* Subject has had previous endovascular repair of the ascending and/or descending thoracic aorta <30 days of implantation of investigational device or previous repair was a non-Medtronic device
* Treatment with the Valiant Mona LSA Thoracic Stent Graft system would require intentional coverage of the left common carotid artery with the stent graft fabric.
* Subject has significant and/or circumferential aortic mural thrombus at either the proximal or distal attachment sites that would compromise fixation and seal of the device.
* Subject is a pregnant female.
* Subject has a known allergy or intolerance to the device components.
* Subject is in acute renal failure or has renal insufficiency with a serum creatinine ≥ 2.0 mg/dL or is on dialysis.
* Subject has a body habitus which prevents adequate visualization of the aorta.
* Subject has coronary artery disease with unstable angina and who has not received treatment.
* Subject has a connective tissue disease (e.g. Marfan's syndrome, medial degeneration).
* Subject has active systemic infection and/or a mycotic aneurysm.
* Subject is currently participating in an investigational drug or device clinical trial that would interfere with the observations of this study.
* Subject has other medical, social, or psychological problems that, in the opinion of the investigator, will interfere with treatment and follow-up procedures.
* Subject has a life expectancy of less than 1 year.
* Subject requires treatment of an infrarenal aneurysm at the time of the implantation.
* Subject has had previous surgical or endovascular treatment of an infra-renal aortic aneurysm <30 days of implantation of investigational device.
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
* Subject has had a cerebral vascular accident (CVA) within 3 months.
* Subject has had a myocardial infarction (MI) within 3 months.
* Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 subjects were enrolled in the study. 30 enrolled subjects were implanted with the study device. The 30-day primary endpoint was evaluated when 29 subjects completed the 30-day follow-up.
Groups:
- Endovascular Repair: Subjects who were appropriate candidates for endovascular repair of the Descending Thoracic Aorta (DTA) who require coverage of the left subclavian artery (LSA) and who met the inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Endovascular Repair
Started | 32
Implanted | 30
Completed | 29
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, Continuous - collected by site
  years | 69.44 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex/Gender - collected by site
  Participants
    Female | 18
    Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Customized - collected by sites
  Participants
    Black or African-American | 5
    Caucasian | 26
    Asian | 1
Region of Enrollment [Number; unit: participants] — Region of Enrollment - collected by site.
  participants
    United States | 32

OUTCOME MEASURES:

1. Primary Outcome: 30 Day Composite Safety Endpoint
Description: Within 1 month (Day 0 - Day 30) from the index procedure, composite endpoint consisting of:
  * Aorta Related Mortality
  * Stroke
  * Paraplegia
  * Left Arm/Hand Ischemia
Time Frame: 1 month
Population: The analysis was performed on all enrolled subjects who were considered evaluable. The subjects were considered enrolled after arterial access is achieved and the Valiant Mona LSA Thoracic Stent Graft System was introduced into the vasculature. Subjects were evaluable if they had the event, or did not have the event and completed a follow-up 15 days or more after the index procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 30
percentage of participants | 10.0 [2.1 to 26.5]

2. Primary Outcome: 30 Day Treatment Success
Description: Treatment success which is defined as technical success (the successful delivery and deployment of the Valiant Mona LSA Thoracic Stent Graft System in the planned location with no unintentional coverage of other vessels, assessed intra-operatively, and the removal of the delivery system) and successful exclusion of the aneurysm or false lumen while maintaining patency of the Main Stent Graft and Branch Stent Graft at 30 day visit. This endpoint is site reported.
Time Frame: 1 month
Population: The analysis was performed on all enrolled subjects who were considered evaluable. There were 3 patients who were not evaluable because they did not have the event and were missing at least one of the three components (technical success, successful exclusion at 30 days, or maintaining patency at the 30 day visit).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 29
percentage of participants | 62.1 [42.3 to 79.3]

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality through 5 years (05DEC2024)
Arm/Group | Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 9/32
Serious Adverse Events (participants affected / at risk) | 30/32
Other Adverse Events (participants affected / at risk) | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Repair (N=32)
Anaemia (Blood and lymphatic system disorders) | 2
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 5
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Coronary Artery Disease (Cardiac disorders) | 1
Coronary Artery Stenosis (Cardiac disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 2
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Chest Pain (General disorders) | 2
Death (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Stent-Graft Endoleak (General disorders) | 3
Sudden Cardiac Death (General disorders) | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1
Transplant Rejection (Immune system disorders) | 1
Appendicitis Perforated (Infections and infestations) | 1
Breast Abscess (Infections and infestations) | 1
Clostridium Difficile Infection (Infections and infestations) | 1
Enterococcal Bacteraemia (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Meningitis Bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Postoperative Wound Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Vascular Access Site Infection (Infections and infestations) | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 2
Arterial Injury (Injury, poisoning and procedural complications) | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 1
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Wound Secretion (Injury, poisoning and procedural complications) | 1
Troponin Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebral Haematoma (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 1
Normal Pressure Hydrocephalus (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional State (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Breast Haematoma (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Lymphadenectomy (Surgical and medical procedures) | 1
Peripheral Endarterectomy (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 1
Aortic Aneurysm (Vascular disorders) | 4
Aortic Aneurysm Rupture (Vascular disorders) | 1
Aortic Dissection (Vascular disorders) | 1
Aortic Dissection Rupture (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive Emergency (Vascular disorders) | 1
Iliac Artery Dissection (Vascular disorders) | 2
Jugular Vein Thrombosis (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
Peripheral Artery Thrombosis (Vascular disorders) | 3
Peripheral Ischaemia (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Peripheral Artery Dissection (Vascular disorders) | 1
Asthenia (General disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Dilated Cardiomyopathy (Cardiac disorders) | 1
Tooth Abscess (Infections and infestations) | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Repair (N=32)
Anaemia (Blood and lymphatic system disorders) | 5
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Angina Unstable (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Atrial Tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac Failure Chronic (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 3
Sinus Bradycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest Pain (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Physical Deconditioning (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Clostridium Difficile Colitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Aortic Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Incision Site Oedema (Injury, poisoning and procedural complications) | 1
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1
Post Procedural Fever (Injury, poisoning and procedural complications) | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1
Postimplantation Syndrome (Injury, poisoning and procedural complications) | 1
Shoulder Fracture (Injury, poisoning and procedural complications) | 1
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 2
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Blood Creatinine Increased (Investigations) | 2
Body Temperature Increased (Investigations) | 1
Peripheral Pulse Decreased (Investigations) | 1
Prostatic Specific Antigen Increased (Investigations) | 1
Transaminases Increased (Investigations) | 1
Urine Output Decreased (Investigations) | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance Disorder (Nervous system disorders) | 1
Bell's Palsy (Nervous system disorders) | 1
Carotid Artery Dissection (Nervous system disorders) | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 1
Taste Disorder (Nervous system disorders) | 1
Thrombosis In Device (Product Issues) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diaphragmatic Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Aneurysm (Vascular disorders) | 2
Aortic Aneurysm (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Hypertensive Urgency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Iliac Artery Dissection (Vascular disorders) | 1
Peripheral Artery Dissection (Vascular disorders) | 1
Subclavian Artery Aneurysm (Vascular disorders) | 1
Subclavian Artery Stenosis (Vascular disorders) | 1
Venous Stenosis (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medtronic owns the data of this clinical study, a single investigation site may access and use the data provided by itself for scientific publications following prior approval by Medtronic.

DOCUMENTS (5):
  • Study Protocol: page 0-50 (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02365467/Prot_000.pdf
  • Study Protocol: 51-100 (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02365467/Prot_001.pdf
  • Study Protocol: 101-150 (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02365467/Prot_002.pdf
  • Study Protocol: 151-200 (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02365467/Prot_003.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02365467/SAP_004.pdf